CLINICAL TRIAL: NCT01428583
Title: A Multicenter, 12-month, Open-label, Single-arm, Safety Study Of Oxycodone Hydrochloride And Naltrexone Hydrochloride Extended-release Capsules In Subjects With Moderate To Severe Chronic Noncancer Pain
Brief Title: Safety Study of Oxycodone Hydrochloride and Naltrexone Hydrochloride Extended-Release Capsules in Subjects With Moderate to Severe Chronic Noncancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Supportive Care
Other Study IDs: ALO-02-10-3001; B4531001 (Other: Alias Study Number)
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Noncancer Pain
Keywords: Chronic noncancer pain; oxycodone; naltrexone
MeSH Terms: interventions — Oxycodone; oxycodone naltrexone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxycodone HCl and naltrexone HCl extended-release capsules (Experimental)
  Interventions: Drug: oxycodone HCl and naltrexone HCl extended-release capsules

INTERVENTIONS:
Drug: oxycodone HCl and naltrexone HCl extended-release capsules — Daily dose range of 20 mg to 160 mg of the oxycodone component in a 24 hour time interval, administered twice daily approximately 12 hours apart (At the discretion of the Investigator, oxycodone HCl and naltrexone HCl extended-release capsules may be administered once daily, at 24 hour intervals.)
  Other Names: ALO-02

SUMMARY:
The study will provide information to assess the benefits versus risks of extended exposure to oxycodone HCl and naltrexone HCl extended-release capsules in a chronic noncancer pain population.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate to severe chronic noncancer pain (duration of at least 3 months) requiring a continuous around-the-clock opioid analgesic for an extended period of time. Conditions may include, but are not limited to, osteoarthritis, chronic low back pain, or other opioid -responsive pain conditions.
* Subject agrees to refrain from taking opioid medications other than study drug during the study. (The exception is during the Pre-Treatment Period when the subject may continue current opioid therapy to guide first 4 weeks of the Treatment Period when the subject may administer immediate-release oxycodone to support conversion to study drug.)

Exclusion Criteria:

* Subject has moderate or severe chronic pain due to cancer, migraine, recent trauma, infection, or other pain expected to be short-term (duration less than 3 months).
* Subject has a documented history of alcohol or drug abuse within 1 year prior to study entry that in the Investigator's judgment would impact subject participation.
* Subject has ongoing or active alcohol or drug abuse that in the Investigator's judgment would impact subject participation.
* Subject has a positive urine drug test for illicit drug use or medications at screening without legitimate medical explanation.
* Subject has a clinically significant medical condition (e.g., cardiovascular, neurological, renal, hepatic, pulmonary, gastrointestinal, endocrine, hematological, immunological, rheumatological, metabolic, or psychiatric) or physical examination, vital signs (VS), 12-lead electrocardiogram (ECG), clinical laboratory abnormalities that in the opinion of the Investigator would impact the safety of the subject during study participation.
* If female, the subject is pregnant or breast-feeding.
* Subject has a known history or known hypersensitivity to oxycodone, oxycodone salts, naltrexone or acetaminophen,or pharmacological similar compounds.
* Subject is historically non-responsive to oxycodone treatment or requires greater than 160 mg oxycodone in a 24-hour time interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (32):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Accord Clinical Research, Port Orange, Florida
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Center for Prospective Outcome Studies, Inc., Atlanta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - Crossroads Research, Owings Mills, Maryland
  - DM Clinical Research, Springfield, Massachusetts
  - MAPS Applied Research Center, Edina, Minnesota
  - Mid-South Anesthesia Consultants, Southaven, Mississippi
  - Healthcare Research, LLC, Hazelwood, Missouri
  - Montana Neuroscience Institute, Missoula, Montana
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Drug Trials America - New York, Hartsdale, New York
  - New York Spine and Wellness Center, North Syracuse, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Center for Clinical Research, LLC - Winston-Salem, Winston-Salem, North Carolina
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Hypothetest, LLC, Roanoke, Virginia

REFERENCES:
- [Derived] Gimbel JS, Rauck RL, Bass A, Wilson J, Pixton G, Malhotra B, Wilson G, Wolfram G. Effects of naltrexone exposure observed in two phase three studies with ALO-02, an extended-release oxycodone surrounding sequestered naltrexone. J Opioid Manag. 2019 Sep/Oct;15(5):417-427. doi: 10.5055/jom.2019.0530. PMID 31849032
- [Derived] Wilson JG, Bass A, Pixton GC, Wolfram G, Rauck RL. Safety and tolerability of ALO-02 (oxycodone hydrochloride and sequestered naltrexone hydrochloride) extended-release capsules in older patients: a pooled analysis of two clinical trials. Curr Med Res Opin. 2020 Jan;36(1):91-99. doi: 10.1080/03007995.2019.1661679. Epub 2019 Sep 17. PMID 31456431
- [Derived] Arora S, Setnik B, Michael D, Hudson JD, Clemmer R, Meisner P, Pixton GC, Goli V, Sommerville KW. A multicenter, 12-month, open-label, single-arm safety study of oxycodone-hydrochloride/naltrexone-hydrochloride extended-release capsules (ALO-02) in patients with moderate-to-severe chronic noncancer pain. J Opioid Manag. 2014 Nov-Dec;10(6):423-36. doi: 10.5055/jom.2014.0239. PMID 25531960
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ALO-02-10-3001&StudyName=Safety%20Study%20of%20Oxycodone%20Hydrochloride%20and%20Naltrexone%20Hydrochloride%20Extended-Release%20Capsules%20in%20Subjects%20With%20Moderate%20to%20Severe%20Chron

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxycodone Hydrochloride (HCl) and Naltrexone HCl: Participants received oxycodone HCl and naltrexone HCl extended-release capsules at an allowable total daily dose range of 20 milligram (mg) oxycodone HCl /2.4 mg naltrexone HCl to 160 mg oxycodone HCl /19.2 mg naltrexone HCl, once daily or twice daily, as per investigators' discretion, for 12 months. Following Month 12, dose might be tapered from the current total daily dose of oxycodone HCl and naltrexone HCl extended-release capsules to the Investigator-determined standard of care based on investigator's discretion.
Period: Overall Study
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Started | 395
Completed | 158
Not Completed | 237
Not completed — Adverse Event | 75
Not completed — Withdrawal by Subject | 51
Not completed — Lack of Efficacy | 37
Not completed — Lost to Follow-up | 17
Not completed — Death | 1
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 12
Not completed — Non-compliant | 25
Not completed — Confirmed positive urine drug test | 8
Not completed — Sponsor's request | 3
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who had at least 1 dose of oxycodone HCl and naltrexone HCl extended-release capsules.
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203
  Male | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Adverse Reactions
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE that was attributed to study drug in a participant who received study drug was defined as an adverse reaction. Treatment-emergent are events between first dose of study drug and up to end of study (2 weeks post-end of month 12) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to end of study (2 weeks post-end of month 12)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
participants
  Adverse event (all causalities) | 343
  Adverse reaction | 207

2. Secondary Outcome: Number of Participants With Treatment Emergent (TE) Adverse Events (AEs) Based on Intensity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Intensity of adverse event was defined on the basis of severity of an event and was classified as; mild (does not interfere with participant's usual function), moderate (interferes to some extent with participant's usual function) and severe (interferes significantly with participant's usual function). Treatment-emergent are events between first dose of study drug and up to end of study (2 weeks post-end of month 12) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to end of study (2 weeks post-end of month 12)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
participants
  Mild | 94
  Moderate | 202
  Severe | 47

3. Secondary Outcome: Percentage of Participants With Clinical Opiate Withdrawal Scale (COWS) Score
Description: The presence and level of clinical opiate withdrawal signs or symptoms was determined by clinician-administered, clinical opiate withdrawal scale (COWS). It contains 11 common opiate withdrawal signs or symptoms rated by clinician (resting pulse rate, gastrointestinal upset, sweating, tremor, restlessness, yawning, pupil size, anxiety or irritability, bone or joint aches, gooseflesh skin, runny nose or tearing), rated on either 3-point, 4-point or 5-point scale, higher score indicated more symptoms of withdrawal. The total score is the sum of all items, ranging from 0 to 48, higher score indicated severe withdrawal. Participants were categorized as less than mild (score 0-4) mild (score 5-12), moderate (score 13-24), moderately severe (score 25-36) or severe (score greater than 36). Percentage of participants with mild (score 5-12), moderate (score 13-24), moderately severe (score 25-36) or severe (score greater than 36) were reported.
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
percentage of participants
  Mild (score 5-12) | 13.2
  Moderate (score 13-24) | 0.0
  Moderately severe (score 25-36) | 0.3
  Severe (score greater than 36) | 0.0

4. Secondary Outcome: Subjective Opiate Withdrawal Scale (SOWS) Score
Description: The presence and level of clinical opiate withdrawal signs or symptoms was determined by participant-reported instrument, subjective opiate withdrawal scale (SOWS). It contains 16 symptoms of opiate withdrawal rated by the participant (anxiety, yawning, sweating, tearing, running nose, goose bumps, shaking, hot flashes, cold flashes, bone or muscle aches, restlessness, nauseous, vomiting, muscle twitch, stomach cramps and feel like using now). Each item is rated on a 5-point scale (0= not at all, 1= a little, 2= moderate, 3= quite a bit, 4= extreme). The total score is the sum of all items, ranging from 0 to 64, higher score indicated severe withdrawal.
Time Frame: Baseline, Week 1, 4, Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: Safety analysis set included all enrolled participants who had at least 1 dose of oxycodone HCl and naltrexone HCl extended-release capsules. Here "n" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
units on a scale
  Baseline (n= 395) | 5.4 (5.49)
  Week 1 (n= 362) | 4.6 (6.15)
  Week 4 (n= 307) | 3.6 (4.32)
  Month 2 (n= 252) | 3.6 (4.70)
  Month 3 (n= 221) | 3.3 (4.53)
  Month 4 (n= 210) | 2.9 (4.30)
  Month 5 (n= 198) | 3.2 (4.56)
  Month 6 (n= 190) | 2.5 (3.27)
  Month 7 (n= 185) | 2.4 (4.07)
  Month 8 (n= 180) | 2.5 (3.74)
  Month 9 (n= 174) | 2.4 (4.08)
  Month 10 (n= 167) | 2.2 (3.25)
  Month 11 (n= 162) | 2.3 (3.53)
  Month 12 (n= 154) | 2.4 (4.09)

5. Other Pre Specified Outcome: Observed Steady-state Plasma Concentrations (Cobs) of Oxycodone
Time Frame: Week 1, 4, Month 2, 3, 6, 9, 12 or early termination
Population: Data was not available to report as PK parameters were plotted by individual participant listings but not summarized for analysis, as per planned analysis.
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Observed Steady-state Plasma Concentrations (Cobs) of Noroxycodone
Description: Noroxycodone was a metabolite of Oxycodone.
Time Frame: Week 1, 4, Month 2, 3, 6, 9, 12 or early termination
Population: as for outcome 5
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Observed Steady-state Plasma Concentrations (Cobs) of Naltrexone
Time Frame: Week 1, 4, Month 2, 3, 6, 9, 12 or early termination
Population: as for outcome 5
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Observed Steady-state Plasma Concentrations (Cobs) of 6-Beta-naltrexol
Description: 6-Beta-naltrexol was a metabolite of naltrexone.
Time Frame: Week 1, 4, Month 2, 3, 6, 9, 12 or early termination
Population: as for outcome 5
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Time to Stabilization of Study Medication
Description: Stabilization was considered to have occurred when: total daily dose of oxycodone and naltrexone remained unchanged for greater than or equal to (>=) 3 consecutive days, daily acetaminophen used remained at 1 gram or less and immediate-release oxycodone was not being used as a rescue medication. Days to stabilization = date of stabilization - date of first dose + 1.
Time Frame: Baseline up to Month 12
Population: Safety analysis set included all enrolled participants who had at least 1 dose of oxycodone HCl and naltrexone HCl extended-release capsules. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: days
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 246
days | 11.0 [3 to 133]

10. Other Pre Specified Outcome: Duration of Exposure to Study Medication
Description: Duration of exposure to study medication during the course of the study was assessed.
Time Frame: Baseline up to 2 weeks after last dose
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
days | 171.0 [1 to 406]

11. Other Pre Specified Outcome: Mean Daily Dose of Study Medication (Oxycodone Component)
Time Frame: Baseline- less than (<) Week 1, Week 1-<4, Week 4-<Month 2, Month 2-<3, Month 3-<4, Month 4-< 5, Month 5-<6, Month 6-<7, Month 7-<8, Month8-<9, Month 9-<10, Month 10-<11, Month 11-<12, Month 12-<End of study (2 weeks post end of Month 12)
Population: Safety analysis set. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: milligram/day
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
milligram/day
  Baseline-less than (<) Week 1 (n= 378) | 38.6 (81.27)
  Week 1-<4 (n= 344) | 51.7 (35.53)
  Week 4-<Month 2 (n= 292) | 62.8 (42.65)
  Month 2-< 3 (n= 238) | 66.1 (40.35)
  Month 3-<4 (n= 217) | 68.0 (40.36)
  Month 4-< 5 (n= 205) | 68.6 (41.49)
  Month 5-<6 (n= 193) | 71.5 (43.58)
  Month 6-<7 (n= 183) | 73.1 (43.22)
  Month 7- <8 (n= 183) | 76.7 (43.76)
  Month 8-<9 (n= 177) | 77.7 (45.67)
  Month 9-<10 (n= 169) | 76.5 (44.58)
  Month 10- <11 (n= 163) | 77.9 (44.45)
  Month 11- <12 (n= 160) | 76.2 (43.14)
  Month 12- <End of study (n= 82) | 26.9 (22.79)

12. Other Pre Specified Outcome: Number of Participants With Rescue Medication (Acetaminophen Tablets)
Description: Participants had acetaminophen up to 2 grams per day during the treatment period of the study as rescue medication.
Time Frame: as for outcome 11
Population: Intent-to-treat (ITT) included all participants in the safety analysis set who had at least 1 pain intensity score reported during treatment. Here "n" signifies those participants who were evaluable at specified time point.
Measure: Number; unit: participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 387
participants
  Baseline-<Week 1 (n= 387) | 256
  Week 1-<4 (n= 361) | 204
  Week 4-<Month 2 (n= 305) | 167
  Month 2-<3 (n= 252) | 124
  Month 3-<4 (n= 222) | 120
  Month 4-<5 (n= 209) | 112
  Month 5-<6 (n= 199) | 104
  Month 6-<7 (n= 191) | 96
  Month 7-<8 (n= 185) | 96
  Month8-<9 (n= 179) | 93
  Month 9-<10 (n= 172) | 79
  Month 10-<11 (n= 167) | 80
  Month 11-<12 (n= 163) | 85
  Month 12-<End of study (n= 95) | 30

13. Other Pre Specified Outcome: Percentage of Participants With Response to Urine Drug Test
Description: Participants with a positive urine drug test for illicit drug substances (marijuana, cocaine, amphetamines, methamphetamines, phencyclidine, and ecstasy), or unexpected drug substances (those other than reported by the participant as therapeutic concomitant medications such as opiates and methadone), or a negative urine test for the expected opioid (oxycodone) was assessed.
Time Frame: Screening, Week 4, Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 or early termination
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
percentage of participants
  Screening (n= 393) | 86.8
  Week 4 (n= 302) | 41.7
  Month 2 (n= 251) | 43.0
  Month 3 (n= 222) | 43.2
  Month 4 (n= 211) | 39.3
  Month 5 (n= 198) | 41.4
  Month 6 (n= 190) | 44.2
  Month 7 (n= 184) | 41.8
  Month 8 (n= 179) | 44.1
  Month 9 (n= 174) | 44.8
  Month 10 (n= 167) | 44.3
  Month 11 (n= 161) | 50.3
  Month 12 or early termination (n= 343) | 57.1

14. Other Pre Specified Outcome: Percentage of Participants With Current Opioid Misuse Measure (COMM) Score of 9 or Above
Description: The COMM is a 17-item self-report questionnaire to monitor for aberrant medication-related behaviors among chronic pain participants. Participants are asked to indicate the frequency of individual behaviors on a scale from 0 to 4 (0 = never, 1 = seldom, 2 = sometimes, 3 = often, 4= very often). The total COMM score is the sum of the 17 item scores with a range from 0 to 68. Higher score indicated a higher risk for aberrant medication- related behavior. A score of 9 or higher was defined as high risk for aberrant medication- related behavior.
Time Frame: Baseline, Week 4, Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 or early termination
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 395
percentage of participants
  Baseline (n= 395) | 21.3
  Week 4 (n= 302) | 8.9
  Month 2 (n= 250) | 10.0
  Month 3 (n= 217) | 8.3
  Month 4 (n= 208) | 6.7
  Month 5 (n= 197) | 5.1
  Month 6 (n= 189) | 2.6
  Month 7 (n= 185) | 3.2
  Month 8 (n= 181) | 5.0
  Month 9 (n= 174) | 5.7
  Month 10 (n= 167) | 4.8
  Month 11 (n= 162) | 3.7
  Month 12 or early termination (n= 333) | 15.3

15. Other Pre Specified Outcome: Mean Daily Dose of Immediate-release Oxycodone as Rescue Medication
Description: Immediate-release oxycodone as a single ingredient product was used as a rescue medication only during the first 4 weeks of the treatment period to support the initiation of oxycodone HCl and naltrexone HCl treatment.
Time Frame: Up to Week 4
Population: Data for mean daily dose of immediate-release oxycodone was not reported because as per protocol and analysis plan it was not planned to be summarized.
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Participants Global Assessment of Treatment Satisfaction
Description: Participant global assessment of treatment satisfaction was scored on a 5-point categorical scale based on response to the question "Please rate your overall satisfaction with the study drug you received?" where 1 = very dissatisfied, 2 = dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = satisfied, 5 = very satisfied.
Time Frame: Week 1, 4, Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, end of treatment
Population: ITT. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 387
unit on a scale
  Week 1 (n= 361) | 3.3 (1.03)
  Week 4 (n= 304) | 3.8 (0.99)
  Month 2 (n= 251) | 3.9 (0.94)
  Month 3 (n= 220) | 4.1 (0.88)
  Month 4 (n= 209) | 4.1 (0.93)
  Month 5 (n= 197) | 4.2 (0.90)
  Month 6 (n= 190) | 4.2 (0.89)
  Month 7 (n= 185) | 4.2 (0.81)
  Month 8 (n= 181) | 4.2 (0.81)
  Month 9 (n= 174) | 4.2 (0.96)
  Month 10 (n= 167) | 4.3 (0.73)
  Month 11 (n= 162) | 4.3 (0.79)
  Month 12 (n= 154) | 4.2 (1.04)
  End of treatment (n= 372) | 3.6 (1.27)

17. Other Pre Specified Outcome: Mean Change From Baseline in Pain Right Now Score at Weeks 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination
Description: The pain intensity scale consisted of 4 questions (pain at its worst in the last 24 hours, pain at its least in the last 24 hours, pain on the average in the last 24 hours and pain right now) each scored on an 11-point numerical rating scale, where 0 = no pain and 10 = pain as bad as you can imagine. "Pain right now" was reported.
Time Frame: Baseline, Week 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination (ET)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 387
units on a scale
  Baseline (n= 386) | 5.6 (2.17)
  Change at Week 1 (n= 360) | -0.6 (2.16)
  Change at Week 4 (n= 306) | -1.3 (2.29)
  Change at Month 2 (n= 251) | -1.6 (2.36)
  Change at Month 3 (n= 218) | -1.7 (2.34)
  Change at Month 4 (n= 208) | -1.8 (2.29)
  Change at Month 5 (n= 197) | -1.8 (2.29)
  Change at Month 6 (n= 189) | -1.8 (2.38)
  Change at Month 7 (n= 184) | -1.7 (2.40)
  Change at Month 8 (n= 180) | -1.8 (2.48)
  Change at Month 9 (n= 172) | -1.8 (2.39)
  Change at Month 10 (n= 166) | -1.7 (2.41)
  Change at Month 11 (n= 161) | -1.9 (2.31)
  Change at Month 12 (n= 153) | -1.9 (2.44)
  Change at Month 12/ET (n= 373) | -1.4 (2.58)

18. Other Pre Specified Outcome: Mean Change From Baseline in Average Pain Score at Weeks 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination
Description: The pain intensity scale consisted of 4 questions (pain at its worst in the last 24 hours, pain at its least in the last 24 hours, pain on the average in the last 24 hours and pain right now) each scored on an 11-point numerical rating scale, where 0 = no pain and 10 = pain as bad as you can imagine. Pain on average in the last 24 hours" was reported.
Time Frame: Baseline, Week 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 387
unit on a scale
  Baseline (n= 384) | 5.9 (1.74)
  Change at Week 1 (n= 357) | -0.6 (1.64)
  Change at Week 4 (n= 303) | -1.2 (1.95)
  Change at Month 2 (n= 250) | -1.5 (2.11)
  Change at Month 3 (n= 219) | -1.7 (2.12)
  Change at Month 4 (n= 206) | -1.7 (2.04)
  Change at Month 5 (n= 196) | -1.7 (2.02)
  Change at Month 6 (n= 189) | -1.7 (2.11)
  Change at Month 7 (n= 184) | -1.7 (2.17)
  Change at Month 8 (n= 180) | -1.9 (2.12)
  Change at Month 9 (n= 173) | -1.8 (2.21)
  Change at Month 10 (n= 166) | -1.7 (2.26)
  Change at Month 11 (n= 161) | -1.8 (2.02)
  Change at Month 12 (n= 153) | -1.9 (2.23)
  Change at Month 12/ET (n= 372) | -1.3 (2.32)

19. Other Pre Specified Outcome: Mean Change From Baseline in Worst Pain Score at Weeks 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination
Description: The pain intensity scale consisted of 4 questions (pain at its worst in the last 24 hours, pain at its least in the last 24 hours, pain on the average in the last 24 hours and pain right now) each scored on an 11-point numerical rating scale, where 0 = no pain and 10 = pain as bad as you can imagine. "Pain at its worst in the last 24 hours" was reported.
Time Frame: Baseline, Week 1, 4, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 12 or Early Termination
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Number analyzed (Participants) | 387
unit on a scale
  Baseline (n= 382) | 7.4 (1.63)
  Change at Week 1 (n= 354) | -0.7 (1.96)
  Change at Week 4 (n= 301) | -1.3 (2.24)
  Change at Month 2 (n= 248) | -1.6 (2.39)
  Change at Month 3 (n= 219) | -1.8 (2.32)
  Change at Month 4 (n= 208) | -1.9 (2.12)
  Change at Month 5 (n= 197) | -1.9 (2.41)
  Change at Month 6 (n= 189) | -2.0 (2.30)
  Change at Month 7 (n= 184) | -2.0 (2.43)
  Change at Month 8 (n= 180) | -2.0 (2.31)
  Change at Month 9 (n= 173) | -2.2 (2.48)
  Change at Month 10 (n= 166) | -2.1 (2.50)
  Change at Month 11 (n= 161) | -2.2 (2.41)
  Change at Month 12 (n= 153) | -2.2 (2.44)
  Change at Month 12/ET (n= 368) | -1.6 (2.52)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Oxycodone Hydrochloride (HCl) and Naltrexone HCl
Serious Adverse Events (participants affected / at risk) | 26/395
Other Adverse Events (participants affected / at risk) | 272/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxycodone Hydrochloride (HCl) and Naltrexone HCl (N=395)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Infected skin ulcer (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Blood pressure increased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxycodone Hydrochloride (HCl) and Naltrexone HCl (N=395)
Nausea (Gastrointestinal disorders) | 100
Constipation (Gastrointestinal disorders) | 84
Vomiting (Gastrointestinal disorders) | 55
Diarrhoea (Gastrointestinal disorders) | 36
Fatigue (General disorders) | 36
Upper respiratory tract infection (Infections and infestations) | 24
Influenza (Infections and infestations) | 20
Back pain (Musculoskeletal and connective tissue disorders) | 25
Headache (Nervous system disorders) | 46
Somnolence (Nervous system disorders) | 37
Dizziness (Nervous system disorders) | 34
Anxiety (Psychiatric disorders) | 30
Insomnia (Psychiatric disorders) | 20
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 24
Pruritus (Skin and subcutaneous tissue disorders) | 21

LIMITATIONS AND CAVEATS:
Outcome measure reporting of Participants With Response to Urine Drug Test were based on qualitative point of contact results only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.